CLINICAL TRIAL: NCT00887731
Title: Clinical Evaluation of a Closed Loop Oxygen Controller for Neonatal Respiratory Care
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: University of Utah (Other)
Responsible Party: Donald Null, University of Utah
Other Study IDs: 30125
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Respiratory Distress Syndrome; Hyperoxia; Prematurity
Keywords: closed loop oxygen controller; premature infants; oxygen exposure
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyperoxia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Part 1 group: Observational study with a convenience sample of ten (10) patients. PART 1 will end when at least 3 of 4 consecutive patients achieve the goal of less than six (6) operator required interruptions per hour for oxygen saturation deviations from study guidelines, or at ten (10) patients.
- Part 2 group: (After successful completion of PART 1) Within patient cross-over study with a randomized cross-over sequence. Sequential data analysis methods will be used to help minimize the patient sample size which will be no more than twenty (20) patients plus up to a maximum of seven (7) who might be eligible from PART 1.
- Part 3 Group: (After successful completion of PART 2) Within patient cross-over study with a randomized cross-over sequence. Studies will last 4 to 12 hours divided in two (2) equal time blocks with one cross-over to either automatic or manual control modes.

SUMMARY:
Nearly forty years ago Berran and coworkers tested an analog oxygen controller to maintain incubator oxygen levels for infants suffering neonatal respiratory disease in order to prevent hyperoxia.

There are at least three clinical issues that this technology addresses: the first is avoidance of episodic hyperoxia; the second is decreasing episodic hypoxia; and the third is lowering cumulative oxygen exposure.

Clinical trials which have used target SpO2 ranging probably help improve all of these problems, but so far there have been no direct measurements of continuous arterial oxygen levels, nor clinical studies which establish the degree to which improving control over blood oxygen saturation decreases the cumulative amount of oxygen exposure. This study will address the later and is an important step in the process of incorporating closed-loop oxygen control technology as a routine standard of neonatal respiratory care.

OBJECTIVES:

PART 1: Test and modify the instruction set for the computerized oxygen controller to achieve a goal of less than six (6) operator required interruptions per hour for oxygen saturation deviations outside of study guidelines.

PART 2: Perform a within patient cross-over trial of the computerized oxygen controller versus standard of care (the patient's care team adjusts the patient's oxygen level) and evaluate the area under the time curve for oxygen exposure between the two control methods.

PART 3:(After successful completion of PART 2) Continuation of the within patient cross-over study with a randomized cross-over sequence. Studies will last 4 to 12 hours divided in two (2) equal time blocks with one cross-over to either automatic or manual control modes. Provision for up to an additional twenty (20) patients to be studied.

DETAILED DESCRIPTION:
Nearly forty years ago Berran and coworkers tested an analog oxygen controller to maintain incubator oxygen levels for infants suffering neonatal respiratory disease in order to prevent hyperoxia.

1. The system was able to regulate to within 1% of the set inspired oxygen level and resulted in stable infant arterial oxygen levels measured transcutaneously. Twenty years later, with the advent of pulse oximetry and computer technology, open loop control of infant oxygen saturation was studied in newborns using computer programs incorporating fuzzy logic and clinical algorithms.
2. During computer-assisted inspired oxygen adjustment there was less variability in pulse oximeter oxygen saturation levels (SpO2) and patients spent more time within the target oxygen saturation range. The next technology step was to move from open to closed loop control, as was done by Claure et al in 2001.
3. These investigators found that closed loop control of inspired oxygen was at least as effective as a fully dedicated nurse in maintaining SpO2 within the target range, and that it may be more effective than a nurse working under routine conditions. Percent of recording time spent at normoxia increased from 66% to 75%. Other bench research suggests that closed loop oxygen controllers based on SpO2 monitoring can have response times within 20 seconds and be able to maintain SpO2 within three percent saturation.
4. In a clinical crossover trial it was shown that compared to routine inspired oxygen control management by bedside personnel, closed loop control of inspired oxygen concentration significantly increased time within target saturation range from 82% to 91%.
5. The importance of controlling oxygen exposure in neonates has been long standing, especially as it relates to retinopathy of prematurity and bronchopulmonary dysplasia. The prospect for decreasing oxygen related morbidities is still a real and an ongoing topic for process change directed to overcoming treatment barriers.
6. Maintaining oxygen saturation tightly within appropriate treatment ranges appears to improve both short and long term outcomes, including developmental indices.
7. Given the improvement in oxygen exposure that can be realized by closed-loop control of inspired oxygen concentration as demonstrated above, the development of commercial devices that incorporate this technology is highly desirable and a positive move toward uniform control of oxygen exposure for neonates. There are at least three clinical issues that this technology addresses: the first is avoidance of episodic hyperoxia; the second is decreasing episodic hypoxia; and the third is lowering cumulative oxygen exposure.

ELIGIBILITY:
Inclusion Criteria:

* Any neonatal intensive care patient who is requiring oxygen therapy as part of their respiratory treatment course will be eligible for this study.
* Parental consent

Exclusion Criteria:

* Infant on room air

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any neonatal intensive care patient who is requiring oxygen therapy as part of their respiratory treatment course will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PART 1: Test and modify the instruction set for the computerized oxygen controller to achieve a goal of less than six (6) operator required interruptions per hour for oxygen saturation deviations outside of study guidelines. | 2-4 hours

SECONDARY OUTCOMES:
PART 2: Perform a within patient cross-over trial of the computerized oxygen controller versus standard of care and evaluate the area under the time curve for oxygen exposure between the two control methods. | 12 hours
Part 3 | 12 hrs
  Perform a within patient cross-over trial of the computerized oxygen controller versus standard of care and evaluate the area under the time curve for oxygen exposure between the two control methods. Studies will last 4 to 12 hours divided in two (2) equal time blocks with one cross-over to either automatic or manual control modes.

CONTACTS AND LOCATIONS:
Overall Officials: Donald N-u-l-l, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah